CLINICAL TRIAL: NCT03973229
Title: The LOW E2 STUDY- Neuroendocrine Risk Mechanisms for Post-traumatic Stress Disorder in Women
Brief Title: Neuroendocrine Risk for PTSD in Women
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Stevens, Assistant Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00103595; 1R01MH117009-01A1 (NIH)
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: PTSD; Trauma
Keywords: Estrogen; Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Stress Disorders, Traumatic | interventions — Ortho Evra

STUDY DESIGN:
Intervention Model Description: Women will participate in one cycle with the estrogen patch and one cycle with the placebo patch. Each cohort will include 40 participants in each of the three study arms for a total of 240 participants.
Who Masked: Participant, Investigator
Masking Description: Randomization will be double blind, with the key held by the study coordinator in a locked file. The study coordinator will do checks of appropriate enrollment to groups after each 20 participants, but no blind will be broken to individuals analyzing study data. Grady pharmacy services will also hold the randomization schedule, as they will dispense the appropriate patch at the appropriate time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Cohort 1: PTSD Receiving Estradiol then Placebo (Experimental): Participants with PTSD will record their first cycle with the Clue app. They will receive the estradiol patch during the second cycle, and the placebo patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch
- Cohort 1: PTSD Receiving Placebo then Estradiol (Experimental): Participants with PTSD will record their first cycle with the Clue app. They will receive the placebo patch during the second cycle, and the estradiol patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch
- Cohort 1: Trauma without PTSD Receiving Estradiol then Placebo (Active Comparator): Participants with trauma exposure will record their first cycle with the Clue app. They will receive the estradiol patch during the second cycle, and the placebo patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch
- Cohort 1: Trauma without PTSD Receiving Placebo then Estradiol (Active Comparator): Participants with trauma exposure will record their first cycle with the Clue app. They will receive the placebo patch during the second cycle, and the estradiol patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch
- Cohort 1: Healthy Controls Receiving Estradiol then Placebo (Active Comparator): Participants without trauma history or psychiatric disorder will record their first cycle with the Clue app. They will receive the estradiol patch during the second cycle, and the placebo patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch
- Cohort 1: Healthy Controls Receiving Placebo then Estradiol (Active Comparator): Participants without trauma history or psychiatric disorder will will record their first cycle with the Clue app. They will receive the placebo patch during the second cycle, and the estradiol patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch
- Cohort 2: PTSD Receiving Estradiol then Placebo (Experimental): Participants with PTSD will begin daily urine ovulation tests on Day 11 of their first cycle, and will record the results with the Clue app. During the second month of cycle monitoring, the MRI will be scheduled 5-7 days after they record a positive ovulation test (during luteal phase) and they will use the estradiol patch before getting the MRI. They will apply the placebo patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch
- Cohort 2: PTSD Receiving Placebo then Estradiol (Experimental): Participants with PTSD will begin daily urine ovulation tests on Day 11 of their first cycle, and will record the results with the Clue app. During the second month of cycle monitoring, the MRI will be scheduled 5-7 days after they record a positive ovulation test (during luteal phase) and they will use the placebo patch before getting the MRI. They will apply the estradiol patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch
- Cohort 2: Trauma Control Receiving Estradiol, then Placebo (Active Comparator): Participants with trauma exposure will begin daily urine ovulation tests on Day 11 of their first cycle, and will record the results with the Clue app. During the second month of cycle monitoring, the MRI will be scheduled 5-7 days after they record a positive ovulation test (during luteal phase) and they will use the estradiol patch before getting the MRI. They will apply the placebo patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch
- Cohort 2: Trauma Control Receiving Placebo then Estradiol (Active Comparator): Participants with trauma exposure will begin daily urine ovulation tests on Day 11 of their first cycle, and will record the results with the Clue app. During the second month of cycle monitoring, the MRI will be scheduled 5-7 days after they record a positive ovulation test (during luteal phase) and they will use the placebo patch before getting the MRI. They will apply the estradiol patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch
- Cohort 2: Healthy Control Receiving Estradiol then Placebo (Active Comparator): Participants without trauma history or psychiatric disorder will begin daily urine ovulation tests on Day 11 of their first cycle, and will record the results with the Clue app. During the second month of cycle monitoring, the MRI will be scheduled 5-7 days after they record a positive ovulation test (during luteal phase) and they will use the estradiol patch before getting the MRI. They will apply the placebo patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch
- Cohort 2: Healthy Control Receiving Placebo then Estradiol (Active Comparator): Participants without trauma history or psychiatric disorder will begin daily urine ovulation tests on Day 11 of their first cycle, and will record the results with the Clue app. During the second month of cycle monitoring, the MRI will be scheduled 5-7 days after they record a positive ovulation test (during luteal phase) and they will use the placebo patch before getting the MRI. They will apply the estradiol patch during the third cycle.
  Interventions: Drug: Estradiol patch; Other: Placebo patch

INTERVENTIONS:
Drug: Estradiol patch — Estradiol (E2) patches at a dose of 100ug will be applied 24-48 hours before the MRI scan is performed.
Other: Placebo patch — Placebo patch identical to the estradiol patch will be applied 24-48 hours before the MRI scan is performed.

SUMMARY:
This study will test for effects of estradiol (E2) on PTSD symptoms and functional magnetic resonance imaging (fMRI) indicators of stress vulnerability, in naturally-cycling women who are not using hormonal birth control. Enrollment will be targeted to create three groups within two cohorts (early follicular phase and luteal phase):

1. PTSD: Women who meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for PTSD
2. Trauma-Exposed (TC): Women matched for age and trauma exposure severity but without PTSD
3. Healthy Control (HC): Women matched for age, but without trauma history or psychiatric disorder (self-reported)

Women will be recruited through Grady Trauma Project (GTP), a large longstanding study of civilian trauma and PTSD conducted at Grady Memorial Hospital in Atlanta, Georgia.

DETAILED DESCRIPTION:
The majority of Americans will experience a traumatic event during their lifetimes. However, women are twice as likely as men to experience negative psychiatric outcomes following trauma, including post-traumatic stress disorder (PTSD) and depression. The reason for the increased prevalence in women is unclear, partially because of the historical lack of investigation of females in both human and pre-clinical animal research. The researchers propose to investigate the role of sex hormones in contributing to women's risk for PTSD. The study will investigate relationships between trauma exposure and women's menstrual cycle, examining key events in the cycle, including menstruation, ovulation, and mood changes. The study will then examine relationships between the level of naturally-cycling estradiol (E2; the primary female sex hormone), and brain-based measures of stress vulnerability. This includes amygdala hyper-reactivity to threat.

The trial will study if trauma-exposed women with lower E2 levels during the luteal phase will report greater PTSD symptoms, and show more stress-vulnerable patterns of brain function. It will also examine the effects of exogenous application of estrogen on PTSD symptoms.

Women will begin tracking their cycle using a free and widely-used cycle-tracking smartphone app "Clue" for one full menstrual cycle.

* For Study Aims 1 & 2 (N=120): Participants will be contacted on the first day of their menstrual period in the second cycle, and scheduled for an MRI with a 4-day window (early follicular phase). Participants will be randomized to begin with either the E2 or placebo patch. The will receive an E2 or placebo patch 1 day prior to the MRI visit, with a blood draw on the morning of the MRI visit (to assess hormone levels), 1 hour prior to scanning. On the first day of the third cycle (onset of menses), women will all be scheduled for their second MRI visit. Participants will experience the opposite condition from their first MRI scan. They will receive an E2 or placebo patch 1 day prior to the MRI visit in the afternoon, with a blood draw on the morning of the MRI visit, 1 hour prior to scanning.
* For Study Aim 3 (N=120): Participants will begin daily urine ovulation tests on Day 11 of their cycle, and will record the results in Clue. When participants record a positive ovulation test during the second month of cycle monitoring, they will be contacted to schedule their MRI visit 5-7 days following ovulation (during the luteal phase). The experimental protocol will otherwise be the same as in Aims 1 and 2, with participants randomized to either E2 or placebo at the first visit and returning the next month for the other condition.

The scientific premise of this study is that low E2 may contribute to stress vulnerability in women. Findings may aid in the development of treatments that will enhance women's mental health outcomes following trauma.

ELIGIBILITY:
Inclusion Criteria:

* African American women
* A menstrual period within the past 60 days
* Able and willing to give informed consent
* Must have a smart phone and willing to install the Clue app

Exclusion Criteria:

* Women currently taking any form of hormone-based birth control or other hormonal supplement
* Women who are pregnant or breastfeeding
* Current psychoactive medication use
* Nicotine use or smoking
* Hypercoagulable conditions
* History of embolism
* Current symptoms of psychosis or bipolar disorder
* History of major head injury or neurological disorder
* Weight >250lbs (a maximum weight to allow for participants to fit comfortably inside the bore of the MRI machine) and typical physical contraindications for MRI such as metal implants

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in amygdala response to fearful faces stimuli | Mid-cycle second cycle, Mid-cycle third cycle (each cycle is an average of 28 days)
  Responses to threat cues will be assessed by fMRI responses as participants view 15 blocks each of fearful face and neutral face stimuli, while amygdala reactivity is measured.
Change in amygdala response to fear conditioning task | Mid-cycle second cycle, Mid-cycle third cycle (each cycle is an average of 28 days)
  Indicators of fear conditioning will be assessed by fMRI during the fear conditioning tasks. Deficits in fear inhibition have been present in persons with PTSD and during phases of the ovarian cycle.
Change in ventromedial prefrontal cortex (vmPFC) activation during the fear extinction task | Mid-cycle second cycle, Mid-cycle third cycle (each cycle is an average of 28 days)
  Indicators of fear extinction will be assessed by fMRI during the fear extinction tasks. Fear extinction is impaired in persons with PTSD and depends on the vmPFC and its inhibition of amygdala responses to threat stimuli.

SECONDARY OUTCOMES:
Change in PTSD checklist for DSM-5 (PCL-5) | Baseline, Mid-cycle second cycle, Mid-cycle third cycle (each cycle is an average of 28 days)
  The severity of self-reported PTSD symptoms will be assessed with the PCL-5. The PCL-5 asks participants to recall the worst stressful event that is currently bothering them the most. Keeping this event in mind, participants respond to 20 questions indicating how bothered they have been by PTSD symptoms. Responses are on a 5-point scale, where 0 = not bothered at all and 4 = extremely bothered. Total raw scores range from 0 to 80 where higher scores indicate greater distress from PTSD symptoms.
Change in Beck Depression Inventory (BDI) | Baseline, Mid-cycle second cycle, Mid-cycle third cycle (each cycle is an average of 28 days)
  The BDI-II is a 21-item instrument assessing depression. Respondents indicate how severe their feelings of depression symptoms are on a scale of 0 (not present) to 3 (most severe). Total raw scores range from 0 to 63, with higher scores indicating greater severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stevens, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
There is an agreement with the National Institute of Mental Health (NIMH) to share deidentified data with Research Domain Criteria (RDoC) database (a centralized NIH database). Raw neuroimaging data and behavioral data for the 3 tasks (Fearful Faces, Fear Conditioning, Fear Extinction), T1 structural brain images, non-identifying demographics, PCL-5, and BDI will be shared.
Supporting Information: Study Protocol
Time Frame: Data will be uploaded to the database every 6 months following the standard NIH schedule (Jan 15 and July 15 of each year of funding). Data will be released publicly within 4 months after submission.
Access Criteria: Data access requests will be submitted to RDoC database, and approved by NIH before data are shared. Only research investigators sponsored by an NIH recognized institution with federal wide assurance will receive access. Any analysis approved by NIH. Web-based access to the RDoC data archive.
URL: https://nda.nih.gov/

DOCUMENTS (1):
  • Informed Consent Form (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT03973229/ICF_000.pdf